CLINICAL TRIAL: NCT05814029
Title: The Effect of Different Mobilization Techniques on Balance, Gait, Jumping and Foot Plantar Pressure in Individuals With Ankle Dorsiflexion Limitation
Brief Title: Different Mobilization Techniques on Balance, Gait, Jumping and Foot Plantar Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammet Ayhan ORAL (Other)
Responsible Party: Sponsor-Investigator, Muhammet Ayhan ORAL, Assist Prof, Kırıkkale University
Organization: Kırıkkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KU-MORAL-001
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Dorsiflexion Deformity of Foot
Keywords: Ankle mobility; Dorsiflexion Limitation; Mobilization with movement; Manuel Therapy; Plantar pressure; Balance; Gait; Jumping
MeSH Terms: interventions — Movement

STUDY DESIGN:
Intervention Model Description: There will be three separate groups in the study. The individuals in the group will be completely different individuals. Each group will receive a different intervention. One of the groups will be the control group
Who Masked: Investigator
Masking Description: Evaluation and mobilization will be performed by two different investigators. The investigator who will make the evaluations will not know in which group the participants are.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The group which mobilization with movement technique applied by clinician (Experimental): 17 individuals in this group, after evaluations, mobilization with movement technique applied by clinician and after that same evaluations will be applied
  Interventions: Other: Mobilization with movement for Ankle
- The group which mobilization with movement technique applied by individual himself (Experimental): 17 individuals in this group, after evaluations, mobilization with movement technique applied by individual himself and after that same evaluations will be applied
  Interventions: Other: Mobilization with movement for Ankle
- Control Group (No Intervention): 16 individuals in this control group, Relevant Extremity will assume a lunge position on a firm mattress with the foot in a weight-bearing stance and the foot in a neutral position. The person will feel uncomfortable and/or the parts will suddenly lunge until the end of their range of motion. No mobilization technique will be applied

INTERVENTIONS:
Other: Mobilization with movement for Ankle — The participant will assume a lunge position on a rigid serving table with the relevant extremity in a weight-bearing stance and the foot in a neutral position. An inelastic belt will be placed around the clinician's waist, flush with the lower edge of the medial malleolus, around the distal tibia and fibula. The clinician will stabilize the talus and forefoot with the web spacing of the hands and pressure dimensions on the talus and forefoot, and maintain posterior to anterior sliding of the tibia over the talus using the arch. The clinician will continue to apply pressure while the person is reporting discomfort and/or while the lunge moves, which will continue until the end of the range of motion. Mobilization will be performed as a 3 set of 10 repetitions.
  Arms: The group which mobilization with movement technique applied by clinician; The group which mobilization with movement technique applied by individual himself

SUMMARY:
Adequate ankle dorsiflexion range of motion is important for normal performance of functional activities such as walking, running and climbing stairs. It is important to gain the ankle dorsiflexion range of motion, which affects the functional activities and sports associated with squats and lunges. Stretching and manual therapy are the most frequently used applications to gain range of motion. Manual therapy has been proposed as a possible treatment to improve mobility and restore arthrokinematics of joints. Movement mobilization, which is a manual therapy method, is an active joint mobilization concept. Talocrural mobilization with the movement technique is an extension of traditional joint mobilizations and allows the patient to engage in therapy in an active, partial weight-bearing lunge position. There are variations of this technique that can be applied by the clinician or by the individual himself. Our aim in this study is to compare the effects of movement and mobilization applications, which can be applied by the clinician or by the individual himself, on balance, gait, jumping and plantar pressure. Healthy asymptomatic individuals between the ages of 18-35 whose active ankle dorsiflexion range of motion as measured by the weight-bearing lunge test in the dominant extremity is below 45˚ will be included in the study. According to the inclusion criteria, the individuals to be included in the study will be randomly divided into three groups. Mobilization technique by the clinician will be applied to one group, and the mobilization technique by the individual himself will be applied to another group. The third group will be the control group. Evaluations will be made before and after mobilization applications. Balance will be evaluated with Y balance test, gait and jump will be evaluated with G-Walk, and plantar pressure will be evaluated with pedobarography device.

DETAILED DESCRIPTION:
Adequate ankle dorsiflexion range of motion is required for normal performance of functional activities such as walking, running, and climbing stairs. Limited ankle dorsiflexion is a common ankle movement disorder that affects squat and lunge-related functional activities and sports. Soft tissue, myofascial tension or muscle tension in the ankle and foot have been identified as the main etiologic factors causing limited ankle dorsiflexion in asymptomatic populations. Limited dorsiflexion range of motion has been associated with genu recurvatum, excessive subtalar joint pronation, ankle sprains, medial tibial stress syndrome, Achilles tendinopathy, plantar fasciitis, anterior knee pain, gastrocnemius strains, and anterior cruciate ligament injuries. Therefore, gaining ankle dorsiflexion range of motion seems to be an important goal in the treatment of lower extremity injuries. Manual therapy has been proposed as a possible treatment to improve mobility and restore arthrokinematics of joints. Movement mobilization is the concept of active joint mobilization. The aim is to render painful movement disorder painless and allow the patient to engage in normal functional activity in the progressive recovery process. Talocrural mobilization with the movement technique is an extension of traditional joint mobilizations and allows the patient to engage in therapy in an active, partial weight-bearing lunge position. There are variations of this technique that can be applied by the clinician or by the individual himself. There are studies showing the effect of clinician-applied motion mobilization on range of motion, static balance, gait, and plantar pressure in different populations. In a study conducted by Reid et al. in individuals with ankle sprains, they observed an increase in ankle dorsiflexion joint range of motion immediately after mobilization with motion for the talocrural joint. In their study, Vicenzino et al. demonstrated the curative effect of motion mobilization techniques on posterior talar shift and dorsiflexion range of motion in individuals with recurrent lateral ankle sprains. Based on this result, they stated that this technique should be considered in rehabilitation programs after lateral ankle sprain. Tomruk et al. showed that the application of the motion mobilization technique to the ankle joint significantly improved postural control in the anteroposterior direction compared to the sham group in healthy individuals. However, overall postural control and dorsiflexion range of motion were significantly increased in both groups compared with initial measurements. On the other hand, the stability limit reaction time was significantly shortened in the motion-only group. In their study, Marrón-Gómez et al. stated that the application of motion mobilization technique and manipulation of the talocrural joint significantly improved ankle dorsiflexion in participants with chronic ankle instability. No significant difference was found between these two techniques, but the results of the application of the motion mobilization technique before the application and the evaluation two days after the application showed larger in-group effect sizes than the high speed and low intensity talocrural joint manipulation. When both treatments were compared with the placebo group, both active interventions were more effective in improving dorsiflexion with larger effect sizes. Yoon et al. reported that passive ankle dorsiflexion improved range of motion, heel-rise time, and dynamic plantar loading during 5-minute walking with a modified motion mobilization technique using talus gliding taping in individuals with limited ankle dorsiflexion. An and Won found that motion ankle mobilization was more effective than simple weight bearing in improving walking speed in stroke patients with limited ankle motion. Gilbreath et al., in their study, showed that there was no significant change in weight-bearing dorsiflexion joint range of motion, in any aspect of the Star Excursion Balance Test, or in Foot and Ankle Ability Measurement-Activities of Daily Living scores after three sessions of motion mobilization technique in individuals with chronic ankle instability. . Although there was no significant change in these parameters, they found a significant improvement in Foot and Ankle Ability Measurement-Sports-Related Activities scores after intervention. Despite these studies investigating the effectiveness of movement mobilization applied by the clinician in different pathologies, there is only one study in the literature comparing the movement applied by the clinician and the individual and the mobilization technique. Stanek and Pieczynski, in their study in healthy individuals with dorsiflexion limitation, stated that both the clinician-applied mobilization and self-mobilization showed significant and sudden increases in the active weight-bearing dorsiflexion joint range of motion when compared to the control group, both while kneeling and standing. They found no significant difference between the groups to which the technique was applied. Based on the findings of this study, clinicians can prescribe self-administered mobilization technique to their patients and expect similar results to clinician-administered mobilization. However, only active dorsiflexion range of motion was evaluated in this study. Although there are studies showing the effect of the movement mobilization technique applied by the clinician on the active dorsiflexion range of motion, foot plantar pressure, jumping and balance, no study has been found in the literature comparing the movements applied by the clinician and the individual in terms of foot plantar pressure, jumping and dynamic balance. Therefore, the aim of this study is to compare the effects of these two techniques in terms of active dorsiflexion range of motion, plantar pressure, jump and dynamic balance in individuals with limited dorsiflexion range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-35
* Volunteering to participate in the study
* Active Dorsiflexion range of motion is below 45˚

Exclusion Criteria:

* Having a history of ankle pain and injury in the last 6 months
* Having a Neurological, Rheumatological or Systemic disease
* Having had any lower extremity surgery

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Active dorsiflexion range of motion (Degree) | 2 Minutes
  Active dorsiflexion range of motion will be evaluated with the Weight Bearing Lunge test. The Weight Bearing Lunge test will be performed using a digital inclinometer. The inclinometer will be placed 15 cm below the anterior part of the tibia and the maximum tibial inclination will be measured while the participant is standing, knee flexed, while transferring weight without lifting the heel off the ground.
Balance (Centimeter) | 10 Minutes
  Y balance test will be used to evaluate the dynamic balance. Participants will be asked to stand barefoot on the weight-bearing platform with their toes positioned back. Then, the participants will be asked to reach anteriorly (ANT), posteromedially (PM), and posterolaterally (PL) three times with their non-weight-bearing extremity.
Gait (second, meter) | 2 Minutes
  Gait analysis will be evaluation with BTS G-WALK device. The G-walk will be placed on the Lumbal 5 level of each participant with the help of a belt. Participants will be asked to walk 8 m at their normal walking speed, turn, and return to their starting point. In this process, the spatiotemporal parameters of the gait will be evaluated.
Jumping (Centimeter) | 3 Minutes
  Jumping performance will be evaluation with BTS G-WALK device. For evaluation, participants will keep their hands on their hips. Three attempts will be made before proceeding to the test. Individuals will be asked to reach the highest possible vertical length with each jump on the dominant leg. Three attempts will be recorded and the average of the jump height and anaerobic performance values for analysis.
Foot Plantar Pressure (centimeter2, contact area %) | 3 Minutes
  Foot plantar pressure will be evaluated using a pedobarographic device. For the measurement, the participants will be asked to stand on the pedobarographic device in a fixed position with bare feet and feet at shoulder level. Participants will be instructed to look across at a fixed point with arms relaxed at both sides. Within the plantar pressure analysis measurements; in static conditions, percentage of contact (%), maximal pressure (N/cm²) and contact area for the dominant foot (cm²), contact surface (%), loads on the fore and hind feet (%) will be determined and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Yusuf DEMIRKAN, Bachelors, Study Chair — Kırıkkale University; Nevin GUZEL, Prof., Study Chair — Gazi University; Gamze COBANOGLU, Master, Study Chair — Gazi University
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marron-Gomez D, Rodriguez-Fernandez AL, Martin-Urrialde JA. The effect of two mobilization techniques on dorsiflexion in people with chronic ankle instability. Phys Ther Sport. 2015 Feb;16(1):10-5. doi: 10.1016/j.ptsp.2014.02.001. Epub 2014 Feb 14. PMID 24679362
- [Background] Hernandez-Guillen D, Roig-Casasus S, Tolsada-Velasco C, Garcia-Gomariz C, Blasco JM. Talus mobilization-based manual therapy is effective for restoring range of motion and enhancing balance in older adults with limited ankle mobility: A randomized controlled trial. Gait Posture. 2022 Mar;93:14-19. doi: 10.1016/j.gaitpost.2022.01.005. Epub 2022 Jan 10. PMID 35042057
- [Background] Brumitt J, Patterson C, Dudley R, Sorenson E, Hill G, Peterson C. COMPARISON of LOWER QUARTER Y-BALANCE TEST SCORES for FEMALE COLLEGIATE VOLLEYBALL PLAYERS BASED on COMPETITION LEVEL, POSITION, and STARTER STATUS. Int J Sports Phys Ther. 2019 Jun;14(3):415-423. doi: 10.26603/ijspt20190415. PMID 31681500
- [Background] Awotidebe TO, Ativie RN, Oke KI, Akindele MO, Adedoyin RA, Olaogun MO, Olubayode TE, Kolawole BA. Relationships among exercise capacity, dynamic balance and gait characteristics of Nigerian patients with type-2 diabetes: an indication for fall prevention. J Exerc Rehabil. 2016 Dec 31;12(6):581-588. doi: 10.12965/jer.1632706.353. eCollection 2016 Dec. PMID 28119881
- [Background] Yazici MV, Cobanoglu G, Yazici G. Test-retest reliability and minimal detectable change for measures of wearable gait analysis system (G-Walk) in children with cerebral palsy. Turk J Med Sci. 2022 Jun;52(3):658-666. doi: 10.55730/1300-0144.5358. Epub 2022 Jun 16. PMID 36326313
- [Background] Rodriguez-Rosell D, Mora-Custodio R, Franco-Marquez F, Yanez-Garcia JM, Gonzalez-Badillo JJ. Traditional vs. Sport-Specific Vertical Jump Tests: Reliability, Validity, and Relationship With the Legs Strength and Sprint Performance in Adult and Teen Soccer and Basketball Players. J Strength Cond Res. 2017 Jan;31(1):196-206. doi: 10.1519/JSC.0000000000001476. PMID 27172267
- [Background] Rabin A, Kozol Z, Spitzer E, Finestone AS. Weight-bearing ankle dorsiflexion range of motion-can side-to-side symmetry be assumed? J Athl Train. 2015 Jan;50(1):30-5. doi: 10.4085/1062-6050-49.3.40. Epub 2014 Oct 20. PMID 25329350
- [Background] Lee J, Park C, Cha Y, You JSH. Comparative effects of different manual techniques on electromyography activity, kinematics, and muscle force in limited ankle dorsiflexion syndrome. J Back Musculoskelet Rehabil. 2021;34(6):1105-1112. doi: 10.3233/BMR-200257. PMID 34057133
- [Background] Hernandez-Guillen D, Blasco JM. A Randomized Controlled Trial Assessing the Evolution of the Weight-Bearing Ankle Dorsiflexion Range of Motion Over 6 Sessions of Talus Mobilizations in Older Adults. Phys Ther. 2020 Apr 17;100(4):645-652. doi: 10.1093/ptj/pzaa003. PMID 31944252
- [Background] Gogate N, Satpute K, Hall T. The effectiveness of mobilization with movement on pain, balance and function following acute and sub acute inversion ankle sprain - A randomized, placebo controlled trial. Phys Ther Sport. 2021 Mar;48:91-100. doi: 10.1016/j.ptsp.2020.12.016. Epub 2020 Dec 23. PMID 33401232
- [Background] An CM, Jo SO. Effects of Talocrural Mobilization with Movement on Ankle Strength, Mobility, and Weight-Bearing Ability in Hemiplegic Patients with Chronic Stroke: A Randomized Controlled Trial. J Stroke Cerebrovasc Dis. 2017 Jan;26(1):169-176. doi: 10.1016/j.jstrokecerebrovasdis.2016.09.005. Epub 2016 Oct 17. PMID 27765557
- [Background] Gilbreath JP, Gaven SL, Van Lunen L, Hoch MC. The effects of mobilization with movement on dorsiflexion range of motion, dynamic balance, and self-reported function in individuals with chronic ankle instability. Man Ther. 2014 Apr;19(2):152-7. doi: 10.1016/j.math.2013.10.001. PMID 24834500
- [Background] Tomruk M, Soysal Tomruk M, Alkan E, Gelecek N. Immediate Effects of Ankle Joint Mobilization With Movement on Postural Control, Range of Motion, and Muscle Strength in Healthy Individuals: A Randomized, Sham-Controlled Trial. J Sport Rehabil. 2020 Nov 1;29(8):1060-1068. doi: 10.1123/jsr.2019-0198. Epub 2019 Nov 19. PMID 31754078
- [Background] Vicenzino B, Branjerdporn M, Teys P, Jordan K. Initial changes in posterior talar glide and dorsiflexion of the ankle after mobilization with movement in individuals with recurrent ankle sprain. J Orthop Sports Phys Ther. 2006 Jul;36(7):464-71. doi: 10.2519/jospt.2006.2265. PMID 16881463
- [Background] Yoon JY, Hwang YI, An DH, Oh JS. Changes in kinetic, kinematic, and temporal parameters of walking in people with limited ankle dorsiflexion: pre-post application of modified mobilization with movement using talus glide taping. J Manipulative Physiol Ther. 2014 Jun;37(5):320-5. doi: 10.1016/j.jmpt.2014.01.007. PMID 24928640
- [Background] An CM, Won JI. Effects of ankle joint mobilization with movement and weight-bearing exercise on knee strength, ankle range of motion, and gait velocity in patients with stroke: a pilot study. J Phys Ther Sci. 2016 Jan;28(2):689-94. doi: 10.1589/jpts.28.689. Epub 2016 Feb 29. PMID 27065565
- [Background] Hall EA, Docherty CL. Validity of clinical outcome measures to evaluate ankle range of motion during the weight-bearing lunge test. J Sci Med Sport. 2017 Jul;20(7):618-621. doi: 10.1016/j.jsams.2016.11.001. Epub 2016 Nov 23. PMID 28108266